CLINICAL TRIAL: NCT06229743
Title: Safety and Effectiveness Study of the Biolinq MicroArray Intradermal Continuous Glucose Biowearable System
Brief Title: Biolinq Safety and Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biolinq Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-011
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Diabetes Mellitus
Keywords: Continuous Glucose Monitoring; Glucose Range Monitoring System
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm (Experimental): All participants will wear at least 1 Biolinq System.
  Interventions: Device: Biolinq System

INTERVENTIONS:
Device: Biolinq System — Participants will wear at least one Biolinq Sensor. The estimated glucose value from the Biolinq Sensor will be compared to a YSI 2300 glucose value from venous blood within a 5 minute window (paired samples).

SUMMARY:
The primary objective of the study is to evaluate the safety and effectiveness of the Biolinq MicroArray Intradermal Continuous Glucose Biowearable System, which is intended to be worn for up to five (5) days (up to 120 hours) in adults with diabetes mellitus (DM). Data collected from this study is intended to be used to support commercial marketing application(s) for the intended commercial patient population of non-insulin-users.

All participants will be asked to wear the Biolinq System and a commercial CGM comparator for five to seven days while taking fingersticks on a commercial Self-Monitoring Blood Glucose Meter. Throughout the sensor wear all participants will come back to the clinic twice for in-clinic days where venous blood draws and fingersticks will be used to compare glucose measurements to a Lab Analyzer (YSI). At the end of sensor wear subjects will return to the clinic to have the sensors removed and then exit the study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 22 years old.
2. Willing and able to provide written signed and dated informed consent.
3. Access to phone or computer with internet to complete subject log.
4. Diagnosis of type 1 diabetes (T1D)/ LADA or type 2 diabetes (T2D) and on intensive insulin therapy (IIT) with known dosing parameters for at least three (3) months prior to the Screening Visit with an A1c of 5.5%-10% or diagnosis of type 2 diabetes (T2D) and on non-intensive insulin therapy (NIIT) or T2D not using insulin with an A1c of 7.5% to 11%.
5. Weigh at least 110 lbs (50 kilograms).
6. Be otherwise in good health, as determined by a medical care professional.
7. Willing to refrain from Acetaminophen use for the duration of study enrollment.
8. If using an automated insulin delivery (AID) system, willing to disable automated features and go into open loop mode during the duration of in-clinic days.

   Device and Glucose Assessments - Willing to:
9. Wear one (1) commercial CGM system on the abdomen per approved labeling and have up to 1 replacement.
10. Wear up to two (2) Biolinq Biowearables simultaneously following the application procedures on the volar forearm for up to 7 days.
11. Participate in two (2) In-Clinic sessions lasting up to 11.5 hours of blood draws (anticipated up to 13 hours on site per visit) each.
12. Perform up to five (5) fingersticks a day with the SMBG device provided during non-in-clinic days.
13. Avoid immersing study devices into water (e.g., no hot tub, SCUBA diving).
14. Wear an activity tracker or record activity levels on a daily log.

Exclusion Criteria:

1. Current participation in another investigational study protocol. (If a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study.) Note: Subjects will not be excluded if enrolled in another observational trial, wherein the subject is in the follow-up phase and no tests/procedures impacting the subject's health are required. Subjects will be excluded if they have been previously enrolled in this study.
2. Work for, are family members with, or live with someone that works for the sponsor or competitor diabetes-related company (includes social media influencers or bloggers).
3. In the investigator's opinion, any reason that may lead to subject non-compliance with study requirements or confound study data.
4. Currently taking Hydroxyurea.
5. Known allergy to medical grade adhesives, acrylic, latex, or isopropyl alcohol.
6. Have dermatological conditions that preclude wearing Biolinq Biowearables (e.g., extensive psoriasis, recent burns, severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, erythema, infection, or other conditions at the discretion of the investigator).
7. For subjects of child-bearing potential, pregnant or not practicing an acceptable form of birth control during the study.
8. Hematocrit measurement via point-of-care (POC) or laboratory testing that is less than the applicable below-mentioned value:

   1. Male: 36.0%
   2. Female: 33.0%
9. Have donated blood, had significant blood loss, or participated in a study with significant blood sampling (340 cc or more) within 56 days prior to study enrollment or plan to participate in such activities during study wear.
10. Required or scheduled to have diathermy, X-ray, MRI, or CT during study wear.
11. In the investigator's opinion, the subject has a history of concomitant medical condition that could interfere with the study participation or present a risk to the safety and welfare of the subject or study staff. Such historical conditions include but are not limited to:

    1. Syncope in past 6 months
    2. Severe hypoglycemia (loss of consciousness, seizure, or emergency medical technician assistance within the past 6 months)
    3. Diabetic ketoacidosis (DKA) requiring hospital admission in the past 6 months
    4. Coagulopathy
    5. Chronic infectious disease (e.g., HIV/AIDS, Hepatitis B or C)
    6. End stage renal disease and currently managed by dialysis or anticipating initiating dialysis during the study wear period
    7. History of congestive heart failure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Advanced Metabolic Care + Research Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Rainier Clinical Research, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was defined as completing the Informed consent process.
Groups:
- Treated Arm: All participants who wore at least 1 Biolinq System.
Period: Overall Study
Arm/Group | Treated Arm
Started | 247
Treated (Primary Sensor) | 202
Left Forearm (Primary Sensor) | 60
Right Forearm (Primary Sensor) | 65
Left Proximal Forearm (Primary Sensor) | 21
Left Distal Forearm (Primary Sensor) | 20
Right Proximal Forearm (Primary Sensor) | 19
Right Distal Forearm (Primary Sensor) | 17
Completed | 190
Not Completed | 57
Not completed — Screen Failure | 45
Not completed — Sensors worn did not meet the revised device specifications | 12

BASELINE CHARACTERISTICS:
Population: 202 participants received at least 1 Biolinq Glucose Sensor. It was pre-specified in the study protocol to report the baseline data for participants irrespective of the number and placement of sensors.
Groups:
- Treated Cohort: All Participants who wore a Biolinq sensor (sensors were blinded and displayed no glucose information to all participants and study personnel).
Arm/Group | Treated Cohort
Number analyzed (Participants) | 202
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 49.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 161
  More than one race | 5
  Unknown or Not Reported | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: In Target Color Indicator - Blue
Description: Number of paired samples of YSI Glucose Readings between 55-207 mg/dL when an unblinded Biolinq sensor would have displayed a blue color indicator (70-180 mg/dL).
Time Frame: 5 days
Population: Performance analysis was limited to the 190 primary sensors to reflect final device specifications. It was pre-specified in the study protocol to report the outcome measures for participants irrespective of the number and placement of sensors, and the data reported in the Outcome Measures are limited to the primary sensor.
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Groups:
- Performance Cohort: 190 participants/sensors that met the final device specifications.
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 7904
Paired Samples - YSI to Biolinq | 7494 [93.3 to 96.0]

2. Primary Outcome: In Target Color Indicator - Yellow
Description: Number of paired samples of YSI Glucose Readings between 154-460 mg/dL when an unblinded Biolinq sensor would have displayed a yellow color indicator (181-400 mg/dL).
Time Frame: 5 days
Population: as for outcome 1
Measure: Count of Units; unit: Paired Samples- YSI to Biolinq
Units Other Than Participants: Paired Samples- YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples- YSI to Biolinq) | 5964
Paired Samples- YSI to Biolinq | 5776 [95.5 to 97.8]

3. Other Pre Specified Outcome: Overall Adverse Device Effect Rate
Description: Overall adverse device effect rate
Time Frame: 5 days
Population: It was pre-specified in the study protocol to report adverse events for participants irrespective of the number and placement of sensors.
Measure: Number; unit: Percentage of Subjects with ADE
Groups:
- Treated Cohort: 202 participants that received at least 1 Biolinq Sensor.
Arm/Group | Treated Cohort
Number analyzed (Participants) | 202
Percentage of Subjects with ADE | 3.5

4. Other Pre Specified Outcome: Individual Adverse Device Effect Rate
Description: Adverse events related to the Biolinq System.
Time Frame: 5 Days
Population: as for outcome 3
Measure: Number; unit: Number of Subjects with ADE
Arm/Group | Treated Cohort
Number analyzed (Participants) | 202
Number of Subjects with ADE
  Pruritus/Itchiness | 2
  Erythema | 2
  Edema | 2
  Ecchymosis/Bruising | 2
  Scabbed Wound | 1

5. Other Pre Specified Outcome: Mean Bias (mg/dL)
Description: Bias is defined by the paired Biolinq Glucose Sensor value minus venous blood sample (YSI) value.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
mg/dL | -7.6 (33.8)

6. Other Pre Specified Outcome: Mean Relative Difference
Description: Relative Difference is defined by the paired Biolinq Glucose Sensor value minus venous blood sample (YSI) value divided by the venous blood sample (YSI) value.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
percentage | -0.7 (19.0)

7. Other Pre Specified Outcome: Type 2 DM Parkes Consensus Error Grid Percentages
Description: The Parkes Error Grid was used to assess the clinical signifiance of blood glucose measurement errors of the Biolinq Glucose Sensor compared to reference values (YSI 2300) by categorizing the errors into risk zones from A-E. The error zone bands were defined in 1994 ADA meeting by a 100 physican survey to assign risk to errors in defined blood glucose ranges then mathmatically calculated to form Zone A-E as described in Parkes et al. Diabetes Care 23:1143-1148, 2000. The outcome measure is the count and percentage of paired samples of Biolinq Glucose Sensor and the YSI 2300 falling into each zone of the pre-defined grid.
Time Frame: 5 days
Population: Performance analysis was limited to the 190 primary sensors to reflect final device specifications. It was pre-specified in the study protocol to report the outcome measures for participants irrespective of the number and placement of sensors, and per protocol the data reported in the Outcome Measures are limited to the primary sensor.
Measure: Count of Units; unit: Errors
Units Other Than Participants: Errors
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Errors) | 13868
Errors
  Zone A- Clinically accurate measurements, no effect on clinical action | 12508
  Zone B - Altered clinical action, little or no effect on clinical outcome | 1339
  C - Altered clinical action, likely to affect clinical outcome | 21
  Zone D - Altered clinical action, could have significant clinical risk | 0
  Zone E - Altered clinical action, could have dangerous consequences | 0

8. Other Pre Specified Outcome: Mean Display Rate
Description: The display rate of the Biolinq Glucose Sensor, which occurs every 5 minutes, is the number of displayable glucose readings (red, blue, and yellow displays) provided divided by the number of expected glucose readings for the given sensor lifetime.
Time Frame: 5 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of displayable readings
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
percentage of displayable readings | 93.9 (13.7)

9. Other Pre Specified Outcome: Median Display Rate
Description: as for outcome 8
Time Frame: 5 days
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: percentage of displayable readings
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
percentage of displayable readings | 98.4 (13.7)

10. Other Pre Specified Outcome: Number of Paired Samples With an Absolute Relative Difference (Between 70-400 mg/dL) Within 20%.
Description: Absolute Relative Difference is defined by the absolute value of Biolinq Glucose Sensor minus venous blood sample (YSI) divided by venous blood sample.
Time Frame: 5 days
Population: as for outcome 7
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 13868
Paired Samples - YSI to Biolinq | 10459

11. Post Hoc Outcome: Number of Paired Samples With Biolinq < 70 mg/dL to YSI Agreement <70 mg/dL, <80 mg/dL, <90 mg/dL, or <100 mg/dL
Description: Number of paired samples of YSI Glucose Readings <70 mg/dL, <80 mg/dL, <90 mg/dL, or <100 mg/dL when an unblinded Biolinq sensor would have displayed a red color indicator (< 70 mg/dL).
Time Frame: 5 days
Population: as for outcome 7
Measure: Number; unit: paired samples - ysi to biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 674
paired samples - ysi to biolinq
  YSI < 70 mg/dL | 498
  YSI < 80 mg/dL | 609
  YSI < 90 mg/dL | 632
  YSI < 100 mg/dL | 649

12. Other Pre Specified Outcome: Number of Paired Samples With an Absolute Relative Difference (Between 70-400 mg/dL) Within 40%
Description: as for outcome 10
Time Frame: 5 days
Population: as for outcome 7
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 13868
Paired Samples - YSI to Biolinq | 13402

13. Other Pre Specified Outcome: Number of Paired Samples With a Day 1 Agreement ± 20%
Description: Agreement is defined by the Biolinq Glucose Sensor minus venous blood sample (YSI) divided by venous blood sample.
Time Frame: Day 1
Population: as for outcome 7
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 4718
Paired Samples - YSI to Biolinq | 3540

14. Other Pre Specified Outcome: Number of Paired Samples With a Day 3 Agreement Within ± 20%
Description: Agreement is defined by the Biolinq Glucose Sensor minus venous blood sample (YSI) divided by venous blood sample.
Time Frame: Day 3
Population: as for outcome 7
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 4730
Paired Samples - YSI to Biolinq | 3521

15. Other Pre Specified Outcome: Number of Paired Samples With a Day 5 Agreement ± 20%
Description: Agreement is defined by the Biolinq Glucose Sensor minus venous blood sample (YSI) divided by venous blood sample.
Time Frame: Day 5
Population: as for outcome 7
Measure: Count of Units; unit: Paired Samples - YSI to Biolinq
Units Other Than Participants: Paired Samples - YSI to Biolinq
Arm/Group | Performance Cohort
Number analyzed (Participants) | 190
Number analyzed (Paired Samples - YSI to Biolinq) | 4420
Paired Samples - YSI to Biolinq | 3398

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow up, up to 7 days.
Description: It was pre-specified in the study protocol to report adverse events for participants irrespective of the number and placement of sensors.
Groups:
- Enrollment Cohort: Participants who signed the Informed Consent.
Arm/Group | Enrollment Cohort
All-Cause Mortality (participants affected / at risk) | 0/247
Serious Adverse Events (participants affected / at risk) | 0/247
Other Adverse Events (participants affected / at risk) | 23/247
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Cohort (N=247)
Headache (Nervous system disorders) | 3 (3)
Pain, IV site (Skin and subcutaneous tissue disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Allergic Reaction (Immune system disorders) | 1 (1)
Ecchymosis/bruising (Vascular disorders) | 4 (4)
Hypoglycemia level 2 (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Irritation/Redness (Skin and subcutaneous tissue disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Pruritus/Itchiness (Skin and subcutaneous tissue disorders) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Edema (Skin and subcutaneous tissue disorders) | 2 (2)
Scabbed Wound (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication before publication of the results from all of the study centers in a peer-reviewed scientific journal or if no article within 12 months after completion of the finalization of the multi-center database. Institution may publish in a peer-reviewed scientific journal. Investigators must provide sponsor with a copy of manuscript 45 days prior to submission for publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT06229743/Prot_SAP_000.pdf